CLINICAL TRIAL: NCT00123227
Title: A Randomised, Double-Blind, Placebo-Controlled, Cardiovascular Magnetic Resonance (CMR) Study to Evaluate the Effect of Rosiglitazone on Carotid Atherosclerotic Plaques in Type 2 Diabetics With Vascular Disease or Hypertension
Brief Title: Rosiglitazone Plaque Study
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Collaborators: GlaxoSmithKline (Industry); CORDA, The Heart Charity (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 02-210
Record Dates: First submitted 2005-07-19; First posted 2005-07-22 (Estimated); Last update posted 2005-08-01 (Estimated); Status verified 2005-05

CONDITIONS: Diabetes Mellitus, Type 2; Vascular Diseases; Hypertension
Keywords: Randomised controlled trial; Rosiglitazone; Cardiovascular magnetic resonance; Diabetes Mellitus; Vascular Diseases; Hypertension
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Vascular Diseases; Hypertension; Diabetes Mellitus | interventions — Rosiglitazone

INTERVENTIONS:
Drug: Rosiglitazone

SUMMARY:
The purpose of this study is to determine whether rosiglitazone, a peroxisome proliferator activated receptor gamma (PPAR-gamma) agonist, induces regression in carotid atherosclerotic plaques in diabetic patients with vascular disease and/or hypertension over a 12 month period.

DETAILED DESCRIPTION:
Rosiglitazone is a new member of the thiazolidinediones (TZDs), a class of drugs which act by binding to peroxisome proliferator activated receptor gamma (PPAR-gamma). It has been suggested that the TZD class od anti-diabetic drug may exhibit anti-atherosclerotic effects. The aim of this study is to evaluate over a 12 month period the potential benefits of rosiglitazone on carotid artery atherosclerotic plaques in the type 2 diabetic population with coexisting vascular disease or hypertension. It is hypothesised that treatment with rosiglitazone will lead to a decrease in plaque size. In addition it is hoped that rosiglitazone will have a positive effect on the plaque composition and stability.

The primary endpoint will be the plaque volume change over 12 months as assessed by cardiovascular magnetic resonance (CMR). The effectiveness of this modality to evaluate the effects of pharmacological agents on atherosclerosis in vivo has been demonstrated in previous studies using statins.

The secondary endpoints will be to define the changes in plaque lipid content, fibrous cap thickness and gadolinium enhancement as a measure of fibrous cap inflammation and plaque neovascularisation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes as defined by the World Health Organization (WHO) criteria
* Male or female patient who is 30 to 75 years of age at screening
* Patients with coexisting vascular disease (previous myocardial infarction, cerebrovascular accident or peripheral vascular disease) or hypertension (BP > 150/90)
* Patients who have initiated statin and fibrate therapy at least 6 months prior to screening, and have been receiving a stable dose for at least 3 months prior to screening. [Note: patients not receiving statin or fibrate therapy will be allowed to enter the study providing that this method of treatment is not required as active treatment for their medical condition at the time of screening; if any of these patients develop the need for statin or fibrate therapy during the course of the study, therapy will be started without the need to withdraw the patient from the study.]
* Female patients must be post-menopausal, surgically sterile, or using effective contraceptive measures. Women of childbearing age must use effective contraceptive measures for at least 1 month prior to visit 1 (screening), and should continue to use the same contraceptive method during the study and for 30 days after discontinuing study treatment.
* Patients who give their signed informed consent to participate.
* Patients with an HbA1c value < 10% at screening visit.
* Patients with evidence of at least one atheromatous plaque causing narrowing of internal carotid artery between 10 and 95%. Diagnosis to be performed prior to randomisation by colour duplex examination.

Exclusion Criteria:

* Patients who have taken >2 concomitant oral anti-hypertensive agents (i.e. oral combination) within the 3 months prior to the screening visit (visit 1)
* Previous exposure to a thiazolidinedione (TZD) or other PPAR-gamma agonist (e.g. rosiglitazone, troglitazone, pioglitazone, GI262570) or participation in a double-blind clinical study involving a TZD or PPAR-gamma agonist where the randomisation code has not been broken prior to visit 1 (screening) of this study.
* Patients who have required the chronic use of insulin for glycaemic control at any time in the past (with the exception of those who have needed short-term insulin use to maintain glycaemic control during a hospitalisation, during pregnancy or during a medical procedure or intervention) or patients with a history of ketoacidosis.
* Use of any investigational drug within 30 days of 5 half-lives preceding the first dose of medication at the start of the study.
* Systolic blood pressure >170 mmHg or diastolic blood pressure > 100mHg.
* Patients with unstable or severe angina or congestive heart failure (New York Heart Association [NYHA] class I-IV)
* History of gangrene or transient ischaemic attack (TIA)
* History of stroke within the previous year.
* Presence of clinically significant hepatic disease (i.e. patients with ALT, total bilirubin, or alkaline phosphatase > 2.5 times the upper limit of the normal laboratory range)
* Any pre-existing condition or clinically significant abnormality identified in the screening (visit 1) physical examination, electrocardiogram, ultrasound examination or laboratory tests which, in the judgement of the investigator, would preclude safe completion of the study.
* Clinically significant anaemia defined by haemoglobin concentration <11g/dL for males, or <10 g/dL for females
* Patients with creatinine > 150 umol/L.
* Women who are lactating, pregnant, or planning to become pregnant during the course of the study.
* Alcohol or drug abuse within the last 6 months.
* Previous surgery to carotid arteries.
* Pacemakers, cerebral aneurysm clips, claustrophobia or any implantable devices incompatible with magnetic resonance imaging.
* Patients exhibiting total occlusion of the internal carotid artery (when assessed by colour duplex examination performed).
* Patients unable to lie supine for 60 minutes.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2002-10; Study Completion 2005-05

PRIMARY OUTCOMES:
Plaque volume change over 12 months as assessed by cardiovascular magnetic resonance (CMR)

SECONDARY OUTCOMES:
Change in plaque lipid content
Change in plaque fibrous cap thickness
Change in plaque gadolinium enhancement as a measure of fibrous cap inflammation and plaque neovascularisation

CONTACTS AND LOCATIONS:
Overall Officials: Dudley J Pennell, MD FRCP FACC, Principal Investigator — Cardiovascular Magnetic Resonance Unit, Royal Brompton Hospital, London UK / National Heart and Lung Institute, Imperial College, London UK
Locations (2):
- United Kingdom (2):
  - Cardiovascular Magnetic Resonance Unit, Royal Brompton Hospital, London
  - St Mary's NHS Trust, London